CLINICAL TRIAL: NCT02615912
Title: A Single-Center, Exploratory Study to Analyze the Dynamics of Skin Microflora Following Exposure to Surfactants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 500-15-0004
Record Dates: First submitted 2015-10-30; First posted 2015-11-26 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis | interventions — sorbitan monopalmitate; Powders; lanpol 5; Sodium Dodecyl Sulfate; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surfactant Exposure (Other): PEG-40 Hydrogenated Castor Oil (Tagat CH40, Evonik) 1.5% Lauryl glucoside (Plantacare® 1200UP, BASF) 1.5% Sorbitan palmitate (SPANTM 40 (powder), Croda) 1.5% Silwet* DA-63 (Momentive) 1.5% Sodium lauryl sulfate (Sigma Aldrich) 1.0% Water
  Interventions: Other: PEG-40 Hydrogenated Castor Oil (Tagat CH40, Evonik) 1.5%; Other: Lauryl glucoside (Plantacare® 1200UP, BASF) 1.5%; Other: Sorbitan palmitate (SPANTM 40 (powder), Croda) 1.5%; Other: Silwet* DA-63 (Momentive) 1.5%; Other: Sodium lauryl sulfate (Sigma Aldrich) 1.0%; Other: Water (control)

INTERVENTIONS:
Other: PEG-40 Hydrogenated Castor Oil (Tagat CH40, Evonik) 1.5%
Other: Lauryl glucoside (Plantacare® 1200UP, BASF) 1.5%
Other: Sorbitan palmitate (SPANTM 40 (powder), Croda) 1.5%
Other: Silwet* DA-63 (Momentive) 1.5%
Other: Sodium lauryl sulfate (Sigma Aldrich) 1.0%
Other: Water (control)

SUMMARY:
The purpose of this study is to understand the changes in skin microflora, skin barrier function, and skin biochemical constituents in response to direct contact with model surfactants used in personal care articles. The results from this study will provide insights into the complex interaction between the skin microbiome and the epidermis after exposure to surfactants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects with Fitzpatrick Skin Types I, II or III

Exclusion Criteria:

* Subjects with visible skin disease, tattoos, skin condition, or abnormal skin color

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Type of microbes present on skin after exposure to various surfactants | 4 days
  Microbes will be identified by metagenomic sequencing
Amount of microbes present on skin after exposure to various surfactants | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Barry Reece, MBA, Principal Investigator — RCTS, Inc.
Locations (1):
- Reliance Clinical Testing Service, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loffler H, Pirker C, Aramaki J, Frosch PJ, Happle R, Effendy I. Evaluation of skin susceptibility to irritancy by routine patch testing with sodium lauryl sulfate. Eur J Dermatol. 2001 Sep-Oct;11(5):416-9. PMID 11525947
- [Background] Hoffman DR, Kroll LM, Basehoar A, Reece B, Cunningham CT, Koenig DW. Immediate and extended effects of sodium lauryl sulphate exposure on stratum corneum natural moisturizing factor. Int J Cosmet Sci. 2014 Feb;36(1):93-101. doi: 10.1111/ics.12101. Epub 2013 Nov 20. PMID 24152302
- [Background] Torma H, Lindberg M, Berne B. Skin barrier disruption by sodium lauryl sulfate-exposure alters the expressions of involucrin, transglutaminase 1, profilaggrin, and kallikreins during the repair phase in human skin in vivo. J Invest Dermatol. 2008 May;128(5):1212-9. doi: 10.1038/sj.jid.5701170. Epub 2007 Nov 15. PMID 18007579
- [Background] Wolcott RD, Gontcharova V, Sun Y, Dowd SE. Evaluation of the bacterial diversity among and within individual venous leg ulcers using bacterial tag-encoded FLX and titanium amplicon pyrosequencing and metagenomic approaches. BMC Microbiol. 2009 Oct 27;9:226. doi: 10.1186/1471-2180-9-226. PMID 19860898
- [Background] Dowd SE, Callaway TR, Wolcott RD, Sun Y, McKeehan T, Hagevoort RG, Edrington TS. Evaluation of the bacterial diversity in the feces of cattle using 16S rDNA bacterial tag-encoded FLX amplicon pyrosequencing (bTEFAP). BMC Microbiol. 2008 Jul 24;8:125. doi: 10.1186/1471-2180-8-125. PMID 18652685
- [Background] Wolcott RD, Dowd SE. A rapid molecular method for characterising bacterial bioburden in chronic wounds. J Wound Care. 2008 Dec;17(12):513-6. doi: 10.12968/jowc.2008.17.12.31769. PMID 19052515